CLINICAL TRIAL: NCT00048711
Title: Open-Label Study of Efficacy and Safety of Recombinant Human N-acetylgalactosamine 4-sulfatase in Patients With MPS VI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASB-01-04
Record Dates: First submitted 2002-11-06; First posted 2002-11-08 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Mucopolysaccharidosis VI
MeSH Terms: conditions — Mucopolysaccharidosis VI | interventions — N-Acetylgalactosamine-4-Sulfatase

INTERVENTIONS:
Drug: N-acetylgalactosamine 4-sulfatase

SUMMARY:
The purpose of the study is evaluate the efficacy, safety, and pharmacokinetics of weekly intravenous infusions of 1 mg/kg recombinant human N-acetylgalactosamine 4-sulfatase (rhASB) in patients diagnosed with Mucopolysaccharidosis VI (MPS VI)

ELIGIBILITY:
Inclusion Criteria:

* Patient consent
* Patient must be five years of age or older
* Patient must have documented biochemical or genetic proof of MPS VI
* Patient must walk at least 1 meter, but less than 250 meters, in the first 6 minutes of the baseline 12-minute walk test
* If female of childbearing potential, patient must have a negative pregnancy test

Exclusion Criteria:

* Patient is under consideration for or has undergone a successful bone marrow transplant (BMT).
* Pregnant or lactating patient
* Patient has received an investigational drug within 30 days prior to study enrollment
* Patient has been previously treated with rhASB
* Patient has a medical condition, serious intercurrent illness, or other extenuating circumstance that may significantly confound study results or decrease study compliance
* Patient has a known hypersensitivity to rhASB or to components of the study drug
* History of cancer (except low grade and fully resolved skin malignancy)

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-03; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
12-minute walk test | weeks 6, 12, 24, 48, 96 and 144
urinary glycoaminoglycan(uGAG)levels | weeks 1, 4, 6, 8, 12

CONTACTS AND LOCATIONS:
Overall Officials: Stuart J Sweidler, MD, Ph.D., Study Director — BioMarin Pharmaceutical
Locations (1):
- BioMarin Pharmaceutical Inc., Novato, California, United States

REFERENCES:
- See also: Related Info — http://www.bmrn.com